CLINICAL TRIAL: NCT06661668
Title: Laparoscopic Implantation of a Gastric Pacemaker is a Low-complication Alternative for Gastroparesis
Brief Title: Laparoscopic Implantation of a Gastric Pacemaker in the Treatment of Gastroparesis
Status: Recruiting | Type: Observational
Sponsor: Evangelic Hospital Kalk Cologne (Other)
Collaborators: Enterra Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Jessica Leers, Prof. Dr. med. Jessica Leers, University of Cologne
Other Study IDs: Gastroparesis_Enterra
Record Dates: First submitted 2024-01-29; First posted 2024-10-28 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-10

CONDITIONS: Gastroparesis; Gastroparesis Postoperative; Gastroparesis Nondiabetic; Gastroparesis With Diabetes Mellitus
Keywords: Gastroparesis; Gastric pacemaker
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Gastroparesis group: Patients scintigraphically proven gastroparesis and failed conservative therapy who undergo laparoscopic gastric pacemaker implantation
  Interventions: Device: Gastric pacemaker (Enterra system) implantation

INTERVENTIONS:
Device: Gastric pacemaker (Enterra system) implantation — Laparascopic implantation of a gastric pacemaker (Enterra system) for patients with therapy refractive gastroparesis

SUMMARY:
Gastroparesis is a burdensome condition that is caused by abnormal motor function of the stomach that results in delayed gastric emptying. It typically manifests with bloating, nausea, vomiting, abdominal pain, and even excessive weight loss and dehydration. The most common causes of gastroparesis are idiopathic, diabetic, medication-induced or iatrogenic (postsurgical) gastroparesis.

Implantation of a gastric neurostimulation device is a surgical option to improve gastric emptying in patients with medication-refractory gastroparesis. Enterra® system is a gastric electrical stimulation that sends mild pulses through leads implanted in the stomach wall that stimulate gastric smooth muscles and nerves in order to improve symptoms and quality of life.

Aim of the investogators' registry trial is to evaluate the feasibility and efficacy of laparoscopic gastric pacemaker implantation for electrical stimulation (Enterra® system). Primary endpoints of the study are symptom severity, health-related quality of life, and frequency of hospitalization before and after pacemaker implantation, perioperative complication rate, and cost effectiveness.

DETAILED DESCRIPTION:
Gastroparesis is a burdensome condition that is caused by abnormal motor function of the stomach that results in delayed gastric emptying. It typically manifests with bloating, nausea, vomiting, abdominal pain, and even excessive weight loss and dehydration. The most common causes of gastroparesis are idiopathic, diabetic, medication-induced or iatrogenic (postsurgical) gastroparesis.

After ruling out mechanical obstruction as an underlying cause of gastroparesis using endoscopy or computed tomography, further assessment includes gastric emptying studies by scintigraphy to confirm the presence of delayed gastric emptying. Severity of symptoms and impact on health-related quality of life can be assessed using the Gastroparesis Cardinal Symptom Index (GCSI) and Gastrointestinal Quality of Life Index (GIQLI).

Management of gastroparesis includes assessment of nutritional status, correction of fluid, electrolytes and nutritional deficiencies, symptomatic therapy, management of the underlying cause of gastroparesis, and improvement of gastric emptying. Implantation of a gastric neurostimulation device is a surgical option to improve gastric emptying in patients with medication-refractory gastroparesis. Enterra® system is a gastric electrical stimulation that sends mild pulses through leads implanted in the stomach wall that stimulate gastric smooth muscles and nerves in order to improve symptoms and quality of life.

Aim of this registry trial is to evaluate the feasibility and efficacy of laparoscopic gastric pacemaker implantation for electrical stimulation (Enterra® system). Primary endpoints of the study are symptom severity, health-related quality of life, and frequency of hospitalization before and after pacemaker implantation, perioperative complication rate, and cost effectiveness.

It is hypothesized that implantation of the Enterra systems leads to a significant improvement of symptoms as well as an increase in health-related quality of life in patients with gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Scintigraphically proven gastroparesis
* Failed conservative therapy
* Severe impairment of quality of life
* Written informed consent
* German language

Exclusion Criteria:

* Age < 18 years
* Prior gastric resection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study includes patients with (1) scintigraphically proven gastroparesis, (2) failed conservative therapy, (3) who undergo laparoscopic gastric pacemaker implantation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms | 5 years
  Symptom severity/Improvement of symptoms pre-/post gastric pacemaker implantation using the standardized Gastroparesis Cardinal Symptom Index (GCSI). The GCSI is based on three subscales: post-prandial fullness/early satiety (4 items); nausea/vomiting (3 items), and bloating (2 items). A total score of 45 can be achieved. A high score indicates more severe symptoms.
Health-related quality of life | 5 years
  Health-related quality of life pre-/post gastric pacemaker implantation using the GIQLI questionnaire (Gastrointestinal Quality of Life Index). GIQLI is a validated instrument to assess HRQoL among patients with gastrointestinal disorders. The questionnaire consists of 36 questions and is subdivided into five subcategories (symptoms, emotion, physical function, social function, and medical treatment). Total scores between 0 and 144 can be achieved. Respective total scores for the specific subcategories are symptoms=76, emotions=20, physical=28, and social=20. Higher scores represent a higher HRQoL.17

SECONDARY OUTCOMES:
Hospital admission | 5 years
  Frequency of hospital admission for further treatment pre/post gastric pacemaker implantation
Perioperative complication rate | 1 year
  Perioperative complications such as wound infection, pain, dysfunctional device

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Leers, Prof., Principal Investigator — Department of Functional Upper GI Surgery
Locations (1):
- Department of Functional Upper GI Surgery, Cologne, North Rhine-Westphalia, Germany